CLINICAL TRIAL: NCT02242487
Title: A 12 Month, Dose-Level Blinded Study Investigating the Safety and Efficacy of CVT 301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena)
Brief Title: Twelve Month Safety and Efficacy Study of CVT-301 In Parkinson's Disease Patients With OFF Episodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVT-301-004E
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Motor fluctuations; levodopa; inhaled drugs; OFF episodes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVT-301 Low Dose (Experimental): Capsules of levodopa inhalational powder used up to 5 times/day for OFF episodes for 12 months duration
  Interventions: Drug: CVT-301
- CVT-301 High Dose (Experimental): Capsules of levodopa inhalational powder used up to 5 times/day for OFF episodes for 12 months duration
  Interventions: Drug: CVT-301

INTERVENTIONS:
Drug: CVT-301
  Other Names: Inhaled levodopa

SUMMARY:
This study is a 12-month, dose-level blinded, multicenter study of 2 inhaled dose levels of CVT-301 for the treatment of up to 5 OFF episodes per day in PD patients experiencing motor fluctuations (OFF episodes). All patients will receive active treatment, but patients will be blinded to dose level. This will serve as an extension to the CVT-301-004 (NCT02240030) study for those patients who participated in that study and remain eligible for this study. In addition, patients who previously completed the CVT-301-003 (NCT01777555), CVT-301-009 (NCT02807675) and CVT-301-005 (NCT02352363) (observational arm completers), as well as CVT-301 naïve patients may be enrolled if they meet the CVT-301-004E eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (PD) diagnosed between the ages of 30 and 80 years;
* Hoehn and Yahr Stage 1-3 in an "on" state;
* Require levodopa-containing medication regimen at least 3 times during the waking day;
* Experience motor fluctuations with a minimum of 2 hours of average daily "off" time per waking day (excluding early morning "off" time) and demonstrate levodopa responsiveness;
* Are on stable PD medication regimen;
* Total daily levodopa (LD) dose <1600 mg/day;
* Able to perform a spirometry maneuver in the ON and OFF states
* Normal cognition confirmed by Mini Mental State Examination (MMSE) score ≥25 ;

Exclusion Criteria:

* Pregnant or lactating females;
* Previous surgery for PD or plan to have stereotactic surgery during the study period. Patients who have had deep brain stimulation [DBS] will also be excluded unless the procedure was performed more than 6 months prior to study enrollment.
* History of psychotic symptoms requiring treatment, or suicide ideation or attempt within last year;
* Known contraindication to the use of levodopa;
* Any significant condition, severe concurrent disease, abnormality or finding that would make patients unsuitable or may compromise patient safety;
* Any any contraindication to performing routine spirometry.

Ages: 30 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (74):
- United States (55):
  - Acorda Site #5020, Scottsdale, Arizona
  - Acorda Site #5042, Fresno, California
  - Acorda Site #5064, Fullerton, California
  - Acorda Site #5035, Loma Linda, California
  - Acorda Site #5027, Long Beach, California
  - Acorda Site #5037, Los Angeles, California
  - Acorda Site #5070, Pasadena, California
  - Acorda Site #5047, Reseda, California
  - Acorda Site #5068, Santa Ana, California
  - Acorda Site #5069, Torrance, California
  - Acorda Site #5052, Washington D.C., District of Columbia
  - Acorda Site #5046, Atlantis, Florida
  - Acorda Site #5053, Aventura, Florida
  - Acorda Site #5013, Boca Raton, Florida
  - Acorda Site #5016, Jacksonville, Florida
  - Acorda Site #5071, Maitland, Florida
  - Acorda Site #5044, Orlando, Florida
  - Acorda Site #5060, Palm Beach Gardens, Florida
  - Acorda Site #5001, Port Charlotte, Florida
  - Acorda Site #5065, St. Petersburg, Florida
  - Acorda Site #5012, Tampa, Florida
  - Acorda Site #5040, Atlanta, Georgia
  - Acorda Site #5025, Chicago, Illinois
  - Acorda Site #5030, Chicago, Illinois
  - Acorda Site #5011, Elk Grove Village, Illinois
  - Acorda Site #5003, Kansas City, Kansas
  - Acorda Site #5067, Baton Rouge, Louisiana
  - Acorda Site #5057, Baltimore, Maryland
  - Acorda Site #5056, Boston, Massachusetts
  - Acorda Site #5018, Boston, Massachusetts
  - Acorda Site #5002, Bingham Farms, Michigan
  - Acorda Site #5014, West Bloomfield, Michigan
  - Acorda Site #5041, Golden Valley, Minnesota
  - Acorda Site #5006, St Louis, Missouri
  - Acorda Site #5023, Las Vegas, Nevada
  - Acorda Site #5028, Albany, New York
  - Acorda Site #5039, Brooklyn, New York
  - Acorda Site #5031, New York, New York
  - Acorda Site #5032, New York, New York
  - Acorda Site #5004, New York, New York
  - Acorda Site #5038, Syracuse, New York
  - Acorda Site #5048, Charlotte, North Carolina
  - Acorda Site #5005, Cleveland, Ohio
  - Acorda Site #5050, Norwood, Ohio
  - Acorda Site #5062, Portland, Oregon
  - Acorda Site #5036, Allentown, Pennsylvania
  - Acorda Site #5010, Philadelphia, Pennsylvania
  - Acorda Site #5058, Willow Grove, Pennsylvania
  - Acorda Site #5022, Charleston, South Carolina
  - Acorda Site #5029, Nashville, Tennessee
  - Acorda Site #5019, Houston, Texas
  - Acorda Site #5045, Houston, Texas
  - Acorda Site #5049, Henrico, Virginia
  - Acorda Site #5059, Virginia Beach, Virginia
  - Acorda Site #5051, Kirkland, Washington
- Canada (3):
  - Acorda Site #5103, London, Ontario
  - Acorda Site #5104, Ottawa, Ontario
  - Acorda Site #5105, Toronto, Ontario
- Czechia (2):
  - Acorda Site #5201, Prague
  - Acorda Site #5203, Prague
- Poland (8):
  - Acorda Site #5305, Gdansk, Zappa
  - Acorda Site #5304, Katowice
  - Acorda Site #5306, Krakow
  - Acorda Site #5303, Krakow
  - Acorda Site #5307, Krakow
  - Acorda Site #5302, Lodz
  - Acorda Site #5308, Warsaw
  - Acorda Site #5301, Warsaw
- Spain (6):
  - Acorda Site #5407, Pamplona, Navarre
  - Acorda Site #5404, Barcelona
  - Acorda Site #5406, Barcelona
  - Acorda Site #5405, Madrid
  - Acorda Site #5403, San Sebastián
  - Acorda Site #5401, Sant Cugat del Vallès

REFERENCES:
- See also: Click here for more information about this study:CVT-301-004E — http://cvt301.acordatrials.com/en/patient/?src=clinicaltrialsgov004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population - Altogether, 325 patients were randomized and 312 patients received at least 1 dose of study drug and were included in the Safety Population. Thirteen patients were randomized but did not receive study drug.
Groups:
- CVT-301 Low Dose: Two capsules of 30 mg each (60 mg total) of levodopa inhalational powder orally inhaled up to 5 times/day for OFF episodes for 12 months duration
  CVT-301
- CVT-301 High Dose: Two capsules of 42 mg each (84 mg total) of levodopa inhalational powder orally inhaled up to 5 times/day for OFF episodes for 12 months duration
  CVT-301
Period: Overall Study
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose
Started | 161 | 164
Completed | 99 | 117
Not Completed | 62 | 47
Not completed — Adverse Event | 13 | 15
Not completed — Lack of Efficacy | 4 | 6
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other - Miscellaneous | 4 | 6
Not completed — Withdrawal by Subject | 37 | 19

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics of 312 is based on the Safety Population of 325 participants randomized less 13 who were randomized and Not Dosed.
Groups:
- CVT-301 Low Dose: 60 mg (two capsules of 30 mg) of levodopa inhalational powder used up to 5 times/day for OFF episodes for 12 months duration
  CVT-301
- CVT-301 High Dose: 84 mg (two capsules of 42 mg) of levodopa inhalational powder used up to 5 times/day for OFF episodes for 12 months duration
  CVT-301
- Total: Total of all reporting groups
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Total
Number analyzed (Participants) | 153 | 159 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 80 | 151
  >=65 years | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.76) | 62.9 (8.34) | 63.4 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 110 | 119 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 3 | 6
  White | 147 | 150 | 297
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 4 | 8
  Czechia | 5 | 3 | 8
  Poland | 39 | 45 | 84
  Spain | 5 | 6 | 11
  United States | 100 | 101 | 201
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.65 (4.820) | 27.59 (4.790) | 27.62 (4.797)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Safety of CVT-301 Change From Baseline for FEV1.
Description: To characterize the effects of CVT-301 on pulmonary safety, as assessed by spirometry FEV1 (forced expiratory volume in 1 second) by treatment group and Treatment Visit (TV). This study was a 12-month, dose-level blinded, multi-center study of 2 inhaled dose levels of CVT-301 for the treatment of up to 5 OFF periods per day in PD (Parkinson's Disease) patients experiencing motor fluctuations (OFF periods). Baseline is defined as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004 study and as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004E study for the rest of the patients.
Time Frame: Change from baseline at 52 weeks
Population: Safety population - Altogether, 325 patients were randomized and 312 patients received at least 1 dose of study drug and were included in the Safety Population. Thirteen patients were randomized but did not receive study drug.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- CVT-301 DL1: 60 mg (two capsules of 30 mg each) of Levodopa Inhalational Powder (LIP) up to 5 times a day.
- CVT-301 DL2: 84 mg (two capsules of 42 mg each) of Levodopa inhalation powder (LIP) up to 5 times a day.
Arm/Group | CVT-301 DL1 | CVT-301 DL2
Number analyzed (Participants) | 153 | 159
Liters
  Baseline | 2.957 (0.6995) | 3.117 (0.7735)
  TV3 (Week 12): number analyzed (Participants) | 141 | 149
  TV3 (Week 12) | -0.059 (0.2321) | -0.078 (0.2108)
  TV4 (Week 24): number analyzed (Participants) | 119 | 136
  TV4 (Week 24) | -0.057 (0.1999) | -0.058 (0.2136)
  TV5 (Week 36): number analyzed (Participants) | 112 | 125
  TV5 (Week 36) | -0.076 (0.2155) | -0.052 (0.2096)
  TV6 (Week 52): number analyzed (Participants) | 105 | 115
  TV6 (Week 52) | -0.086 (0.2238) | -0.097 (0.2230)

2. Primary Outcome: Pulmonary Safety for CVT-301 Change From Baseline for FVC.
Description: To characterize the effects of CVT-301 on pulmonary safety, as assessed by spirometry FVC, (forced vital capacity) by treatment group and Treatment Visit (TV). This study was a 12-month, dose-level blinded, multi-center study of 2 inhaled dose levels of CVT-301 for the treatment of up to 5 OFF periods per day in PD patients experiencing motor fluctuations (OFF periods). Baseline is defined as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004 study and as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004E study for the rest of the patients.
Time Frame: Change from baseline at 52 weeks
Population: Safety Population - Safety population - Altogether, 325 patients were randomized and 312 patients received at least 1 dose of study drug and were included in the Safety Population. Thirteen patients were randomized but did not receive study drug.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | CVT-301 DL1 | CVT-301 DL2
Number analyzed (Participants) | 153 | 159
Liter
  Baseline | 3.840 (0.9047) | 4.045 (0.9811)
  TV3 (Week 12): number analyzed (Participants) | 141 | 149
  TV3 (Week 12) | -0.064 (0.2575) | -0.086 (0.2667)
  TV4 (Week 24): number analyzed (Participants) | 119 | 136
  TV4 (Week 24) | -0.053 (0.2710) | -0.062 (0.2688)
  TV5 (Week 36): number analyzed (Participants) | 112 | 125
  TV5 (Week 36) | -0.089 (0.3051) | -0.050 (0.2659)
  TV6 (Week 52): number analyzed (Participants) | 105 | 115
  TV6 (Week 52) | -0.106 (0.2866) | -0.089 (0.2747)

3. Primary Outcome: Pulmonary Safety for CVT-301 Change From Baseline for (FEV1/FVC).
Description: To characterize the effects of CVT-301 on pulmonary safety, as assessed by spirometry FEV1/FVC (FEV1-forced expiratory volume in 1 second and (FVC) forced vital capacity ratio) by treatment group and Treatment Visit (TV). This study was a 12-month, dose-level blinded, multi-center study of 2 inhaled dose levels of CVT-301 for the treatment of up to 5 OFF periods per day in PD (Parkinson's Disease) patients experiencing motor fluctuations (OFF periods). Baseline is defined as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004 study and as the last non-missing assessment before the first dose of CVT-301 in CVT-301-004E study for the rest of the patients.
Time Frame: Change from baseline at 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio %
Arm/Group | CVT-301 DL1 | CVT-301 DL2
Number analyzed (Participants) | 153 | 159
Ratio %
  Baseline | 77.2 (5.24) | 77.2 (6.00)
  TV3 (Week 12): number analyzed (Participants) | 141 | 149
  TV3 (Week 12) | -0.2 (3.35) | -0.3 (2.89)
  TV4 (Week 24): number analyzed (Participants) | 119 | 136
  TV4 (Week 24) | -0.3 (3.64) | -0.3 (2.91)
  TV5 (Week 36): number analyzed (Participants) | 112 | 125
  TV5 (Week 36) | -0.3 (2.75) | -0.3 (3.02)
  TV6 (Week 52): number analyzed (Participants) | 105 | 115
  TV6 (Week 52) | -0.2 (3.36) | -0.7 (3.51)

4. Secondary Outcome: Count of Patients Achieving Resolution of an OFF to an ON State Within 60 Minutes.
Description: Count of patients achieving resolution of an OFF to an ON state within 60 minutes after study drug is administered in the clinic, and maintaining the ON state at 60 minutes after study drug administration (per the examiner's subjective assessment).
Time Frame: At Treatment Visit - TV6 (Week 52)
Population: ITT (Intent-to-Treat) Population
Measure: Count of Participants; unit: Participants
Arm/Group | CVT-301 DL1 | CVT-301 DL2
Number analyzed (Participants) | 144 | 153
Participants | 78 | 92

5. Secondary Outcome: Change From Baseline in OFF Time.
Description: Patient reported total daily OFF time and was assessed by the patient and recorded in the patient Diary. An "OFF state" is defined as the time when medication is not providing benefit with respect to mobility, slowness, and stiffness. OFF episodes may be heralded by non-motor symptoms (e.g., pain, anxiety) prior to the appearance of motor symptoms. Patients will record their ON and OFF states in their diaries at home.
Time Frame: Change from baseline through 12 months duration of outpatient use
Population: ITT - (Intent-to-Treat) Population. Patients who discontinue the study prior to a treatment visit are not included in the analysis for that treatment visit. Therefore, the number of patients decreases with each successive treatment visit.
Measure: Least Squares Mean (Standard Error); unit: Hours
Groups:
- CVT-301 DL1: 60 mg (two capsules of 30 mg each) of Levodopa Inhalation Powder (LIP)
- CVT-301 DL2: 84 mg (two capsules of 42 mg each) of Levodopa inhalation powder (LIP)
Arm/Group | CVT-301 DL1 | CVT-301 DL2
Number analyzed (Participants) | 144 | 153
Hours
  TV2 (Week 4): number analyzed (Participants) | 137 | 143
  TV2 (Week 4) | -0.33 (0.221) | -0.55 (0.217)
  TV3 (Week 12): number analyzed (Participants) | 133 | 139
  TV3 (Week 12) | -0.23 (0.232) | -0.38 (0.227)
  TV4 (Week 24): number analyzed (Participants) | 114 | 130
  TV4 (Week 24) | -0.65 (0.235) | -0.73 (0.227)
  TV5 (Week 36): number analyzed (Participants) | 102 | 116
  TV5 (Week 36) | -0.49 (0.238) | -0.92 (0.230)
  TV6 (Week 52): number analyzed (Participants) | 94 | 110
  TV6 (Week 52) | -0.70 (0.239) | -0.88 (0.229)

ADVERSE EVENTS:
Time Frame: 12-month period
Groups:
- CVT-301 Low Dose: 60 mg (two capsules of 30 mg each) of Levodopa Inhalational Powder (LIP) up to 5 times a day for OFF episodes for 12 months duration.
- CVT-301 HIgh Dose: 84 mg (two capsules of 42 mg each) of Levodopa inhalation powder (LIP) up to 5 times a day for OFF episodes for 12 months duration.
Arm/Group | CVT-301 Low Dose | CVT-301 HIgh Dose
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/159
Serious Adverse Events (participants affected / at risk) | 22/153 | 13/159
Other Adverse Events (participants affected / at risk) | 81/153 | 69/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVT-301 Low Dose (N=153) | CVT-301 HIgh Dose (N=159)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Mycardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Naseau (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomititng (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Prostrate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostrate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device connection tissue (Product Issues) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide threat (Psychiatric disorders) | 0 (0) | 1 (1)
Bone graft (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVT-301 Low Dose (N=153) | CVT-301 HIgh Dose (N=159)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 23 (27)
Fall (Injury, poisoning and procedural complications) | 24 (26) | 17 (22)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 12 (13)
Nasopharyngitis (Infections and infestations) | 8 (8) | 4 (5)
Dyskinesia (Nervous system disorders) | 6 (6) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT02242487/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02242487/SAP_001.pdf